CLINICAL TRIAL: NCT02853578
Title: National Clinical Study, Multicentric, Single Arm to Evaluate the Efficacy and Safety of Busonid® (Budesonide 200 mcg and 400 mcg) to Treat Asthma Not Controlled or Partially Controlled
Brief Title: Busonid® (Budesonide 200 mcg and 400 mcg) to Treat Asthma Not Controlled or Partially Controlled
Acronym: Laennec
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: The viability of the study is being analyzed
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACH-BSN-03(14/14)
Record Dates: First submitted 2016-07-25; First posted 2016-08-03 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Busonid (budesonide 200mcg and 400mcg) (Experimental): It´s a capsule with inhalatoin powder composed of budesonide 200mcg or 400mcg. The experimental drug will be dispensed in a cartridge containing 60 capsules of 200 mcg or 400 mcg and an inhaler. It should be stored at room temperature (between 15 and 30°C) and protected from moisture.
  Regarding the dosage, the 80 study participants will perform an inhalation 200mcg every 12 hours (400 mcg / day). During follow-up visits (V1 and V2) the attending physician will assess the need for increased PSI dose to 400 mcg every 12 hours (800mcg / day). Study participants should rinse the mouth with water and / or brush your teeth immediately after use of the drug.
  The duration of treatment may be 12 weeks.
  Interventions: Drug: Busonid (budesonide 200mcg and 400mcg)

INTERVENTIONS:
Drug: Busonid (budesonide 200mcg and 400mcg) — cartridge containing 60 tablets of 200 mcg or 400 mcg and an inhaler;
  1 application (inhalation) of 200mcg every 12 noon (400 mcg / day). During the visits of monitoring (V1 and V2) the doctor in charge assess the need to increase the dose of PSI 400mcg for every 12 hours (800mcg / day); treatment for 12 weeks.
  Other Names: Busonid

SUMMARY:
National clinical trial, phase III, multicenter, single-arm, efficacy study, 80 participants of both sexes, aged equal or more than 12 and less than 65 years. The group will use Busonid® (budesonide 200mcg and 400mcg) one application (inhalation) of 200 mcg every 12 hours (400mcg / day). During follow-up visits if the participant has not shown an increase in forced expiratory volume in one second greater than 12% and greater than 0,20L or 200ml in spirometry compared with baseline visit, will increase the dose to 800 mcg / day (2x 400 mcg day).

The study aims to revalidate by the National Health Surveillance Agency (ANVISA) the registration of the drug Busonid® which there is a vast scientific literature on the pre-clinical and clinical evidence that the efficacy and safety of budesonide. Thus, outlined is a single-arm study, which is applied to the study of the group of participants the same intervention for a certain period and the participants are evaluated for response.

DETAILED DESCRIPTION:
Busonid® is composed of budesonide and has two performances of 200mcg and 400mcg. It is a corticosteroid hormone with topical anti-inflammatory activity. The slow and continuous release of budesonide in the airways due to their esterification and their short plasma half life increases the selectivity of the corticosteroid to the airways, in patients with asthma, inhaled corticosteroids have a broad spectrum of anti-inflammatory effects, such as reducing the number of inflammatory cells in the lungs and inhibiting the synthesis and release of cytokines and other inflammatory mediators.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled asthma diagnosis or partially controlled in according to the Guidelines of the Brazilian Society of Pneumology and Phlebology for Asthma Management - 2012;
* Capacity of survey participants or legal guardians to understand and consent to the participation of the research participant in this clinical study, expressed by signing the informed consent form;
* Ability of children survey participants 18 years understand and nod their participation in this clinical study, manifested by signing the informed assent form;
* Baseline forced expiratory volume in one second in screening visit between 55% and 85% of predicted value (before bronchodilator use), including the extremes (ensuring that the lung function test has been performed properly);
* Increase of 12% and 200 ml of forced expiratory volume in one second after the reversibility test at screening visit / initiation of treatment.

Exclusion Criteria:

* Diagnosis of pneumonia, pneumothorax, pneumomediastinum, COPD, pulmonary tuberculosis, deficiency α1anti antitrypsin, lung mycosis (blastomycosis, histoplasmosis), bronchiectasis, pulmonary cystic fibrosis or other significant respiratory disease, according to the investigator;
* Pneumothorax history, pulmonary tuberculosis, lung mycosis (blastomycosis, histoplasmosis) and COPD;
* Immunosuppressive therapy;
* Survey participants with immunosuppression of any kind;
* Thoracic surgery history or any prior neoplastic process of the lung;
* Significant heart disease;
* Four or more systemic corticosteroid courses in the last 12 months;
* Participants who have needed hospitalization or care in the emergency room or emergency service (duration> 12 hours) to airway obstruction control (for exacerbation of asthma), at least once within the last three (03) months;
* History of asthma crisis with risk of death;
* Ventilatory support needs due to respiratory failure secondary to asthma within the past five (05) years;
* Infection of the upper respiratory tract or lower (viral or bacterial) within the last four (04) weeks prior to study entry;
* Any finding of clinical observation (clinical evaluation / physical) that is interpreted by the medical researcher as a risk to the research participant in the clinical study;
* Known hypersensitivity to drug components used during the study;
* Use of forbidden drugs in the clinical study described in Protocol;
* Smokers and former smokers;
* HIV infection, whether on antiretroviral treatment;
* History of abuse of illicit drugs;
* Disorders diagnosis of hypothalamic-pituitary-adrenal axis (hypocortisolism or hypercortisolism);
* Presence of severe obstruction of lung airflow that may present a risk of death;
* Women in reproductive age who do not agree to use hormonal or barrier methods of contraception; except the participants declared that they perform sexual practices or exercise them not to reproductive form;
* Female participants in a period of pregnancy or breastfeeding;
* Clinical trial protocols of participation in the last twelve (12) months (CNS Resolution 251 of August 7, 1997, Part III, sub-item J), unless the investigator considers that there may be a direct benefit to it;
* Family relationship to the second degree or bond with employees or employees of Sponsor and Research Center.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Busonid® (budesonide 200 mcg and 400 mcg) in the treatment of asthma after the initiation of treatment (FEV1) | 12 weeks
  The absolute change in forced expiratory volume in one second [FEV1 (L)], 12 weeks after start of treatment (VF) compared to baseline (V0) was measured by spirometry test.

SECONDARY OUTCOMES:
Evaluate the FEV1 (L) during treatment compared to baseline. | 4, 8 and 12 weeks
  Absolute change of FEV1 (L) during treatment (weeks 4, 8 and 12) compared to baseline (week 0).
Evaluate the FEV1 (% of predicted) during treatment compared to baseline. | 4, 8 and 12 weeks
  Absolute change of FEV1 (% of predicted) during treatment (weeks 4, 8 and 12) compared to baseline (week 0).
Evaluate the FEV1 / FVC during treatment compared to baseline. | 4, 8 and 12 weeks
  Absolute change of FEV1 / FVC during treatment (weeks 4, 8 and 12) compared to baseline (week 0).
Evaluate the peak expiratory flow behavior measured each morning and evening throughout the treatment as compared to baseline. | 2, 4, 6, 8, 10 and 12 weeks
  Absolute variation in peak expiratory flow, measured in the morning and evening, through the peak expiratory flow meter laptop at weeks 2, 4, 6, 8, 10 and 12 relative to baseline morning and evening, which will be measured on the day of V0. The peak expiratory flow of weeks 2, 4, 6, 8, 10 and 12 will be determined by the arithmetic mean of the last seven days prior to the week in review.
Evaluate the occurrence of nighttime awakenings due to symptoms asthma during treatment. | 12 weeks
  Nights rate with awakenings due to asthma symptoms, set at 2-week intervals (1 and 2; 3 and 4; 5 and 6; 7 and 8; 9 and 10; 11 and 12), as assessed by daily participant.
Assess the need for use of rescue medication over treatment. | 12 weeks
  Average number of rescue medication used by jets day set at 2 week intervals (1 and 2; 3 and 4; 5 and 6; 7 and 8; 9 and 10; 11 and 12) as daily participant.
Assess satisfaction to treatment by the investigator and participant search / legal representative throughout the treatment. | 4, 8 and 12 weeks
  Satisfaction with treatment, according to investigator assessment and the research participant / legal representative, expressed by the Visual Analogue Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Elie Fiss, Principal Investigator — Multidisciplinary Studies Center CEPES of the ABC Medical School
Locations (5):
- Brazil (5):
  - Centro de Estudos Multidisciplinar CEPES da Faculdade de Medicina do ABC, Santo André, São Paulo
  - Centro de Pesquisa do Hospital Nipo Brasileiro, São Paulo
  - Centro de Pesquisa em Pneumologia da Santa Casa de São Paulo, São Paulo
  - Centro Paulista de Investigação Clínica - CEPIC, São Paulo
  - IMA Brasil - Instituto de Medicina Avançada, São Paulo